CLINICAL TRIAL: NCT00976885
Title: Oxygen Consumption Required by Stroke Patients During Completion of the Modified Rivermead Mobility Index (MRMI)
Status: Completed | Type: Observational
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Alice YM Jones, The Hong Kong Polytechnic University
Other Study IDs: HSEARS20090209006
Record Dates: First submitted 2009-09-14; First posted 2009-09-15 (Estimated); Last update posted 2009-09-15 (Estimated); Status verified 2009-09

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional

GROUPS / COHORTS (2):
- Subjects with normal health
- Subjects with Stroke

SUMMARY:
The aim of this study was to measure the oxygen consumption and peak heart rate achieved during Modified Rivermead Mobility Index (MRMI) assessment in age-matched, healthy and stroke patients, and assess the efficacy of the MRMI tasks for aerobic training in patients with stroke.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of hemisphere stroke
* aged fifty or above
* ambulatory with/ without walking aid
* had ability to provide informed consent and understand the evaluation procedures

Exclusion Criteria:

* brainstem and cerebellar lesion
* unconscious or drowsy
* musculoskeletal, respiratory or other disease that may limit activity of daily livings
* serious cardiovascular disease

Min Age: 50 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: stroke unit of local hospital and community groups
Sampling Method: Non-Probability Sample

PRIMARY OUTCOMES:
Oxygen consumption

CONTACTS AND LOCATIONS:
Locations (1):
- Cardiopulmonary and exercise physiology laboratory, The Hong Kong Polytechnic University, Hong Kong, China